CLINICAL TRIAL: NCT04428255
Title: A Randomized, Double-blind, Placebo-controlled, Phase 2/3 Operational Seamless Designed Clinical Study to Evaluate the Efficacy and Safety of HBM9161 Weekly Subcutaneous Injection in Patients With Primary Immune Thrombocytopenia
Brief Title: A Clinical Study on the Efficacy and Safety of HBM9161 in Patients With ITP
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Harbour BioMed (Guangzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 9161.4
Record Dates: First submitted 2020-06-09; First posted 2020-06-11 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Primary Immune Thrombocytopenic Purpura
Keywords: ITP

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HBM9161 Dose A (Experimental): Patients will be randomized in a 1:1:1 ratio to HBM9161 (Dose A or Dose B) or placebo
  Interventions: Drug: HBM9161 Dose A
- HBM9161 Dose B (Experimental): Patients will be randomized in a 1:1:1 ratio to HBM9161 (Dose A or Dose B) or placebo
  Interventions: Drug: HBM9161 Dose B
- Placebo (Placebo Comparator): Patients will be randomized in a 1:1:1 ratio to HBM9161 (Dose A or Dose B) or placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HBM9161 Dose A — HBM9161 (Dose A or Dose B) or matching placebo will be administered IV weekly
  Arms: HBM9161 Dose A
Drug: HBM9161 Dose B — HBM9161 (Dose A or Dose B) or matching placebo will be administered IV weekly
  Arms: HBM9161 Dose B
Drug: Placebo — HBM9161 (Dose A or Dose B) or matching placebo will be administered IV weekly
  Arms: Placebo

SUMMARY:
To select a dose and to make a decision for Phase 3 study

DETAILED DESCRIPTION:
The onset of primary immune thrombocytopenia is thought to be increased platelet destruction and decreased platelet production due to anti-platelet antibodies. HBM9161 is a fully human anti-FcRn monoclonal antibody that can effectively remove pathogenic IgG, thereby relieving platelet destruction and rapidly increasing platelet counts in patients. The study will be conducted in a Phase 2/3 operational seamless design, with group Dose A and Dose B of HBM9161 and a placebo group in Phase 2.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age at the screening visit, male or female.
2. Persistent or chronic ITP whose average number of platelet at the screening visit and pre-dose (at least 1 day apart) is < 30 × 10^9/L, and not > 35 × 10^9/L for any of two tests. No severe bleeding within 4 weeks prior to the screening visit.
3. Patients who have received and failed at least 1 first line of ITP therapy (glucocorticoids and/or intravenous gamma globulin), or who are contraindicated, intolerable, or refuse standard therapy.
4. Patients will be allowed to use a stable dose of concomitant drugs for the treatment of ITP. e.g., glucocorticoid, danazol, immunosuppressant (azathioprine, cyclosporine A, mycophenolate mofetil) and eltrombopag.

Exclusion Criteria:

1. Other autoimmune systemic diseases other than ITP.
2. Multi-lineage immune cytopenias, such as Evan's syndrome, autoimmune pancytopenia.
3. Secondary ITP.
4. Received a vaccine within 4 weeks prior to the first dose of the study drug or planned during the study.
5. Use of anticoagulants or any agents that have antiplatelet effect or can affect thrombopoiesis within 3 weeks prior to the first dose of the study drug.
6. Received blood transfusion within 1 week prior to the first dose of the study drug.
7. Received the intravenous gamma globulin, anti-D immunoglobulin, or plasmapheresis within 2 weeks prior to the first dose of the study drug.
8. Received high-dose dexamethasone or high-dose methylprednisolone within 2 weeks prior to the first dose of the study drug.
9. Received recombinant human thrombopoietin (rhTPO) within 4 weeks prior to the first does of the study drug.
10. Received rituximab or other non-rituximab anti-CD20 drugs within 6 months prior to the first does of the study drug.
11. Treated with splenectomy within 4 weeks prior to first dose of the study drug.
12. Any thromboembolic or embolic events within 12 months prior to the first does of the study drug.
13. Serum total IgG < 700 mg/dL at the screening visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2020-07-21 (Actual); Primary Completion 2021-07-17 (Estimated); Study Completion 2023-03-11 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who achieve the early response. | 7 weeks
  The primary endpoint of phase 2

SECONDARY OUTCOMES:
Proportion of patients who achieve platelet count ≥ 50 × 10^9/L at least 2 times within 7 weeks. | 7 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Renchi Yang, Principal Investigator — Hematology hospital, Chinese academy of medical sciences
Locations (1):
- Hematology hospital, Chinese academy of medical sciences, Tianjin, Tianjin Municipality, China

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-27): https://cdn.clinicaltrials.gov/large-docs/55/NCT04428255/Prot_SAP_000.pdf